CLINICAL TRIAL: NCT01889745
Title: A Phase I Clinical Study, Randomized, Single-blind,Placebo-controlled, Multiple Doses, Dose Escalation Study fo the Safety, Tolerability and Pharmacokinetics of HX-1171 in Healthy Male Subjects.
Brief Title: A Phase I Clinical Study of the Safety, Tolerability and Pharmacokinetics of HX-1171 in Healthy Male Subjects.
Acronym: HX-1171
Status: Temporarily not available | Type: Expanded Access
Sponsor: Biotoxtech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013_0361
Record Dates: First submitted 2013-06-20; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
MeSH Terms: interventions — 1-O-hexyl-2,3,5-trimethylhydroquinone

INTERVENTIONS:
Drug: HX-1171 — Anti-oxidatant, Anti-inflamation
  Other Names: 1-O-hexyl-2,3,5-trimethylhydroquinone; HX-1171 500mg

SUMMARY:
This study is designed to multiple dose and dose escalation study

DETAILED DESCRIPTION:
A Phase I Clinical Study, Randomized, Single-blind, Placebo-controlled, Single Dose Escalation Study of the Safety, Tolerabiluty, and Pharmacokinetics of HX-1171 in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 20 to 40 years at screening.
* Be able to comply with the requirement of the study. Subject must provide written informed consent prior to study participation.

Exclusion Criteria:

* History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or gastrointestinal disorders.
* History of known hypersensitivity to drugs including HX-1171.

Ages: 20 Years to 40 Years | Sex: Male
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Special City of Seoul, South Korea

REFERENCES:
- See also: Asan medical center — http://ctc.amc.seoul.kr